CLINICAL TRIAL: NCT06337643
Title: A Phase 1, First-in Human, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study of the Tolerability, Safety, and Immunogenicity of MVX01, a Pneumococcal Vaccine Candidate, in Healthy Adult Participants
Brief Title: A Study to Evaluate Tolerability, Safety and Immunogenicity of MVX01 Pneumococcal Vaccine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Matrivax Research and Development Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: MVX01-01
Record Dates: First submitted 2023-03-20; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Pneumococcal Vaccine
Keywords: Streptococcus Pneumoniae Infection; Pneumonia; S. pneumoniae; Pneumonia, Bacterial; Healthy Human
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia; Pneumonia, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Cohort 1 is open-label. Cohorts 2-5 include two open-label sentinel participants each and the remainder of the participants are randomized and double-blind to either MVX01 or MVX01 Placebo (Participant & Site).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MVX01 Vaccine - Cohort 1 (Experimental): MVX01 Vaccine: liquid formulation, 0.5 mL intramuscular injection, 10 μg Frequency: 2 doses administered approximately 1 month apart Age: 18-50 years,
  Interventions: Biological: MVX01
- MVX01 Vaccine or Placebo - Cohort 2 (Experimental): MVX01 Vaccine: liquid formulation, 0.5 mL intramuscular injection, 30 μg, or Placebo: liquid formulation, 0.5 mL intramuscular injection Frequency: 2 doses administered approximately 1 month apart Age: 18-50 years
  Interventions: Biological: MVX01; Biological: MVX01 Placebo
- MVX01 Vaccine or Placebo - Cohort 3 (Experimental): MVX01 Vaccine: liquid formulation, 0.5 mL intramuscular injection, 60 μg, or Placebo: liquid formulation, 0.5 mL intramuscular injection Frequency: 2 doses administered approximately 1 month apart Age: 18-50 years
  Interventions: Biological: MVX01; Biological: MVX01 Placebo
- MVX01 Vaccine or Placebo - Cohort 4 (Experimental): MVX01 Vaccine: liquid formulation, 0.5 mL intramuscular injection, 90 μg, or Placebo: liquid formulation, 0.5 mL intramuscular injection Frequency: 2 doses administered approximately 1 month apart Age: 18-50 years
  Interventions: Biological: MVX01; Biological: MVX01 Placebo
- MVX01 Vaccine or Placebo - Cohort 5 (Experimental): MVX01 Vaccine: liquid formulation, 0.5 mL intramuscular injection, 90 μg, or Placebo: liquid formulation, 0.5 mL intramuscular injection Frequency: 2 doses administered approximately 1 month apart Age: 60-75 years
  Interventions: Biological: MVX01; Biological: MVX01 Placebo

INTERVENTIONS:
Biological: MVX01 — Pneumococcal Vaccine Candidate
Biological: MVX01 Placebo — Placebo
  Arms: MVX01 Vaccine or Placebo - Cohort 2; MVX01 Vaccine or Placebo - Cohort 3; MVX01 Vaccine or Placebo - Cohort 4; MVX01 Vaccine or Placebo - Cohort 5

SUMMARY:
The objectives of this first-in-human study is to evaluate the tolerability, safety, and immunogenicity of MVX01, a pneumococcal vaccine candidate, at four dose levels.

DETAILED DESCRIPTION:
The study will enroll five cohorts. Ascending doses of MVX01 will be evaluated in cohorts 1-4, in participants 18-50 years of age. The highest tolerated dose from cohorts 1-4 will be evaluated in cohort 5, in participants 60-75 years of age. Cohort 1 will be open-label. Cohorts 2-5 will enroll two open-label sentinel participants followed by the remainder of the cohort which will be randomized and double-blind. Each participant will be administered two doses of study intervention via intramuscular injection, approximately 1 month apart. Immunogenicity will be evaluated up to approximately 6 months following administration of the second dose.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be male or non-pregnant, non-lactating female ≥ 18 to ≤ 50 years of age for Cohorts 1 to 4 and ≥ 60 to ≤ 75 years of age for Cohort 5, at the time of signing the informed consent.
* Body mass index within the range 18 to 32 kg/m2 (inclusive) for Cohorts 1-4. Body mass index within the range 18 to 35 kg/m2 (inclusive) for Cohort 5.
* Participants who are free of clinically significant acute or chronic health conditions in the opinion of the Investigator.
* Have provided written informed consent prior to screening procedures.
* Participant's screening laboratory test results must be either within the normal range or deemed as not clinically significant by the Investigator.
* Venous access considered adequate for collection of safety laboratory samples and immunogenicity samples.
* Contraceptive use by males and females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. In addition, women of childbearing potential must agree to avoid heterosexual activity for a period of 14 days prior to the administration of study intervention.

Exclusion Criteria:

* Positive screening test suggesting a current infection due to human immunodeficiency virus, hepatitis C virus, or hepatitis B virus infection.
* Symptoms of active respiratory illness at the time of the first dose of study intervention or close contact with a known SARS-CoV-2 positive patient within 10 days of first dose of study intervention.
* Suspected or known alcohol and/or illicit drug abuse within the past 5 years.
* Regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Electrocardiogram abnormalities outside of accepted ranges (with some exceptions) or results considered to be clinically significant. Participants with QT interval corrected for heart rate according to Fridericia's formula > 450 msec (if male) or > 460 msec (if female) will be excluded.
* History of confirmed pneumococcal infection based on participant report of medical history during the previous 12 months.
* Use of any investigational (non-registered) drug within 30 days or 5 half-lives of the investigational drug prior to receiving the first dose of study intervention. All investigational (non-registered) drugs used should be noted.
* Use of chronic immunosuppressant agents or other immune-modifying drugs within 6 months prior to receiving the first dose of study intervention. Short-term use of corticosteroids (< 14 days) for an acute illness are allowed but last dose should be ≥ 28 days prior to administration of the first dose of study intervention. The use of topical, inhaled, and nasal glucocorticoids is permitted.
* Receipt of immunoglobulins and/or any blood products within the 3 months preceding Day 1 or planned administration of such products during the study and up Visit 6 (Day 57 [± 4 days]).
* Is planning to become pregnant in the time period from Screening up to 30 days following the last dose of study intervention.
* History of allergic disease, neurologic disease, or untoward reactions likely to be exacerbated by any component of the vaccine and/or known hypersensitivity to any component of the vaccine.
* Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with evaluation of the study intervention or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
* Known or suspected severe immunological dysfunction in the opinion of the Investigator.
* History of administration of any vaccine within 30 days of prior to receiving the first dose of study intervention. Should a vaccine have been administered within the 30-day timeframe, inclusion into the study will be at the discretion of the Investigator. Vaccines may not be administered until after Visit 6 (Day 57 [± 4 days]). Participants should not intend to receive a licensed pneumococcal vaccine until after Visit 7 (Day 210 [± 14 days]). Participants will not be excluded based on previously having received a licensed pneumococcal vaccine as long as it was administered at least 30 days prior to receiving the first dose of study intervention.
* Unwilling or unable to forego donation of sperm, egg, blood, plasma, or platelets from Screening through Visit 6 (Day 57 [± 4 days]).
* In the opinion of the Investigator, any participant with a physical or laboratory finding or past medical history that might suggest a good quality of life for the participant is likely to be < 24 months at the time of Screening examination.
* Participants who, in the opinion of the Investigator, will not be able to comply with all the study procedures and visits as outlined in the protocol, including follow-up.
* A staff member or family member of a staff member of the clinical research organization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-04-16 (Estimated); Study Completion 2024-04-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of immediate reactogenicity adverse events | Up to 30 minutes after each dose
  Number and percentage of immediate reactogenicity events by severity.
  Including:
  * Local expected at injection site: erythema/redness; induration/hardening; pain; pruritus/itching; tenderness.
  * Systemic expected: fatigue; fever; flu-like symptoms; headache; myalgia/muscle pain; nausea; rash; vomiting.
Incidence of solicited reactogenicity events | Up to 7 days after each dose
  Number and percentage of solicited reactogenicity adverse events by severity.
  Including:
  * Local expected at injection site: erythema/redness; induration/hardening; pain; pruritus/itching; tenderness.
  * Systemic expected: fatigue; fever; flu-like symptoms; headache; myalgia/muscle pain; nausea; rash; vomiting
Incidence of adverse events (AEs) | Up to study day 61
  Number and percentage of adverse events reported spontaneously by the participant.
  The following summaries are planned:
  * Overview of TEAEs.
  * All TEAEs.events.
  * All TEAEs by relationship to study intervention.
  * All TEAEs leading to discontinuation.
  * All TEAEs leading to death.
  * All TEAEs by severity.
Incidence of Serious Adverse Events (SAEs) and New-Onset Chronic Illness (NOCI) | Up to study day 224
  Number and percentage of serious adverse events and new-onset chronic illnesses as determined by discretion of the investigator.
  The following summaries are planned:
  * SAEs/NOCIs throughout study).
  * All SAEs considered at least possibly related to study intervention.
Changes in safety laboratory results compared to baseline | Up to study day 61
  Assessment of adverse changes from baseline in safety laboratory results (standard panels for hematology, blood chemistry and urinalysis) that meet criteria as an adverse event as described in "Guidance for Industry Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, FDA 2007".
Changes in vital signs compared to baseline | Up to study day 61
  Assessment of changes in vital signs (SBP, DBP, HR, RR, oral body temp) that meet criteria as an adverse event as described in "Guidance for Industry Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, FDA 2007".
Geometric Mean Titer (GMT) post immunization of Anti-pneumolysin (PLY) and anti-choline binding protein A (CbpA) | Up to study day 224
  Anti-pneumolysin and anti-choline binding protein A serum immunoglobulin G antibody geometric mean titer as measured by enzyme-linked immunosorbent assay (ELISA) compared baseline.
  The anti-PLY and anti-CbpA antibody titers will be measured as >=2- and >=4-fold above baseline to determine GMTs and rates of seroconversion.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Velocity (Meridian) Clinical Research, Savannah, Georgia
  - Alliance for Multispecialty Research (AMR), Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No